CLINICAL TRIAL: NCT03611114
Title: Effects of Blood Orange Juice Consumption on Endothelial Function in Healthy Overweight/Obese Men and Premenopausal Women of European Origin
Brief Title: The Impact of Citrus Products on Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Karen Birch, PhD, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BIOSCI 15-030
Record Dates: First submitted 2018-04-18; First posted 2018-08-02 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Healthy; Overweight and Obesity
Keywords: endothelial function; flow mediated dilation; lipid profile; blood pressure; flavanones; Caucasian
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood orange juice (Experimental): Subjects will be asked to consume blood orange juice (400 ml/day) for 2 weeks.
  Interventions: Dietary Supplement: Blood orange juice
- Control drink (Placebo Comparator): Subjects will be asked to consume a control drink (400 ml/day) for 2 weeks.
  Interventions: Dietary Supplement: Control drink

INTERVENTIONS:
Dietary Supplement: Blood orange juice
  Arms: Blood orange juice
Dietary Supplement: Control drink
  Arms: Control drink

SUMMARY:
Epidemiological studies have indicated that the consumption of citrus fruit is inversely associated with the risk of cardiovascular disease. However, clinical data regarding the effects of blood orange juice upon endothelial function is scarce. This randomised, crossover study investigates whether blood orange juice compared to a control drink improves blood vessel function and other cardiovascular health indicators (such as blood pressure and blood lipids). All the subjects will be asked to consume blood orange juice and a control drink in a randomised order, each over a 2-week period, divided by a 1-week wash out period.

DETAILED DESCRIPTION:
Endothelial function measured via flow mediated dilation (FMD), blood pressure, anthropometric measures, lipid profile, high-sensitivity C-reactive protein (hsCRP) and endothelin 1 (ET-1), cyclic guanosine monophosphate (cGMP) will be evaluated in healthy overweight/obese Caucasians prior to and following 2-week consumption of blood orange juice and a control drink. Evaluation of endothelial function as measured by FMD will be conducted on specific days of the menstrual cycle to minimise the fluctuation in oestrogen levels in premenopausal women, which will be monitored in serum samples.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Caucasians (of European origin)
* BMI > 25 kg/m2

Exclusion Criteria:

* Presence of cardiovascular diseases
* Smoking
* Use of medications or dietary supplements (vitamins, antioxidants)
* On a special diet and/or a training program to change weight

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in flow mediated dilation between baseline and endpoint within the intervention group vs. control group | Baseline and 2 weeks; after 1-week wash out, another baseline and 2 weeks.
  FMD will be evaluated prior to and following 2-week consumption of either blood orange juice or a control drink.

SECONDARY OUTCOMES:
Changes in blood pressure between baseline and endpoint within the intervention group vs. control group | Baseline and 2 weeks; after 1-week wash out, another baseline and 2 weeks.
  Blood pressure will be measured prior to and following 2-week consumption of either blood orange juice or a control drink.
Changes in lipid profile between baseline and endpoint within the intervention group vs. control group | Baseline and 2 weeks; after 1-week wash out, another baseline and 2 weeks.
  Serum total cholesterol, HDL cholesterol, LDL cholesterol will be measured prior to and following 2-week consumption of either blood orange juice or a control drink.
Changes in high sensitivity C-reactive protein between baseline and endpoint within the intervention group vs. control group | Baseline and 2 weeks; after 1-week wash out, another baseline and 2 weeks.
  Serum hsCRP will be measured prior to and following 2-week consumption of either blood orange juice or a control drink.
Changes in endothelin-1 (ET-1) between baseline and endpoint within the intervention group vs. control group | Baseline and 2 weeks; after 1-week wash out, another baseline and 2 weeks.
  Serum ET-1 will be measured prior to and following 2-week consumption of either blood orange juice or a control drink.
Changes in oestradiol between baseline and endpoint within the intervention group vs. control group | Baseline and 2 weeks; after 1-week wash out, another baseline and 2 weeks.
  Serum oestradiol will be measured prior to and following 2-week consumption of either blood orange juice or a control drink.
Changes in flavanone metabolites between baseline and endpoint within the intervention group vs. control group | Baseline and 2 weeks; after 1-week wash out, another baseline and 2 weeks.
  Flavanone metabolites will be measured prior to and following 2-week consumption of either blood orange juice or a control drink.
Changes in cyclic guanosine monophosphate (cGMP) between baseline and endpoint within the intervention group vs. control group | Baseline and 2 weeks; after 1-week wash out, another baseline and 2 weeks.
  Cyclic guanosine monophosphate (cGMP) will be measured prior to and following 2-week consumption of either blood orange juice or a control drink.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Li, PhD, Principal Investigator — University of Leeds; Karen M Birch, PhD, Study Director — University of Leeds; Christine Bosch, PhD, Study Chair — University of Leeds
Locations (1):
- University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller-Delp JM, Lubahn DB, Nichol KE, Philips BJ, Price EM, Curran EM, Laughlin MH. Regulation of nitric oxide-dependent vasodilation in coronary arteries of estrogen receptor-alpha-deficient mice. Am J Physiol Heart Circ Physiol. 2003 Nov;285(5):H2150-7. doi: 10.1152/ajpheart.00966.2002. Epub 2003 Jul 24. PMID 12881205
- [Background] Perticone F, Ceravolo R, Candigliota M, Ventura G, Iacopino S, Sinopoli F, Mattioli PL. Obesity and body fat distribution induce endothelial dysfunction by oxidative stress: protective effect of vitamin C. Diabetes. 2001 Jan;50(1):159-65. doi: 10.2337/diabetes.50.1.159. PMID 11147782
- [Background] Thijssen DH, Black MA, Pyke KE, Padilla J, Atkinson G, Harris RA, Parker B, Widlansky ME, Tschakovsky ME, Green DJ. Assessment of flow-mediated dilation in humans: a methodological and physiological guideline. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H2-12. doi: 10.1152/ajpheart.00471.2010. Epub 2010 Oct 15. PMID 20952670
- [Derived] Li L, Lyall GK, Martinez-Blazquez JA, Vallejo F, A Tomas-Barberan F, Birch KM, Boesch C. Blood Orange Juice Consumption Increases Flow-Mediated Dilation in Adults with Overweight and Obesity: A Randomized Controlled Trial. J Nutr. 2020 Sep 1;150(9):2287-2294. doi: 10.1093/jn/nxaa158. PMID 32510144

DOCUMENTS (2):
  • Study Protocol (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03611114/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03611114/SAP_001.pdf